CLINICAL TRIAL: NCT03489876
Title: Comparison of Synthetic Cartilage Implant Versus Osteochondral Autologous Transfer for Advanced Hallux Rigidus, A Prospective Randomized Controlled Clinical Trial
Brief Title: Synthetic Cartilage Implant vs Osteochondral Autograft Transfer for Advanced 1st Metatarsal Phalangeal Joint Arthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient enrollment.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SynCartImp_Amin
Record Dates: First submitted 2018-03-19; First posted 2018-04-06 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Metatarsophalangeal Joint Arthritis
Keywords: Metatarsophalangeal Joint; Arthritis; Synthetic Cartilage Implant; Cartiva; Osteochondral Autograft Transfer
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Intervention Model Description: Upon eligibility verification and informed consent, computer-based randomization will allot patients into one of the two treatment groups, either synthetic cartilage implant or osteochondral autograft transfer.
Masking Description: The computer-based randomization sequence will be concealed from investigators using REDCap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Synthetic Cartilage Implant (Experimental): Participants receive the synthetic cartilage implant. The synthetic cartilage implant that will be used is the Cartiva implant.
  Interventions: Device: Synthetic Cartilage Implant
- Osteochondral Autograft Transfer (Active Comparator): Participants receive the current standard osteochondral autograft transfer procedure.
  Interventions: Procedure: Osteochondral Autograft Transfer

INTERVENTIONS:
Device: Synthetic Cartilage Implant — The Synthetic Cartilage Implant will be implanted in to the first metatarsal head according to the manufacturer's recommendations.
  Other Names: Cartiva
  Arms: Synthetic Cartilage Implant
Procedure: Osteochondral Autograft Transfer — The osteochondral autograft transfer will be harvested from the ipsilateral lateral femoral condyle (or contralateral if a previous ipsilateral total knee anthroplasty or trauma) and the graft will be transferred to the first metatarsal head.
  Arms: Osteochondral Autograft Transfer

SUMMARY:
This is a prospective, randomized, controlled clinical trial comparing synthetic cartilage implantation versus osteochondral autograft transfer for treatment of first metatarsophalangeal (MTP) arthritis. This data will allow for accurate comparisons between the two groups in regards to functional outcome, clinical outcome, pain relief, and complications.

DETAILED DESCRIPTION:
First MTP joint arthritis or hallux rigidus is the most common arthritic condition of the foot. Historically, there have been several options to treat this condition surgically, but the current standard for advanced hallux rigidus is first MTP anthrodesis. Newer joint preserving procedures offer patients effective relief of pain and improving functional outcomes as well as maintaining, and potentially improving, range of motion for the first MTP joint. Osteochondral autograft transfer has been shown to be an effective treatment for hallux rigidus, and involves harvesting a small cylindrical osteochondral graft from a site remote of the first MTP joint and transferring the graft to the head of the first metatarsal. A new synthetic cartilage implant, Cartiva, has been shown to have equivalent functional outcomes, pain scores, and complications to anthrodesis, but the first MTP range of motion in the Cartiva group was maintained or even improved in some patients.

This is a prospective, randomized, controlled clinical trial comparing synthetic cartilage implantation versus osteochondral autograft transfer for treatment of first metatarsophalangeal (MTP) arthritis. The hypothesis is that clinical range of motion, pain scores, subjective clinical outcomes, and complications will not be clinically inferior with the synthetic cartilage implant group compared to the osteochondral autograft transfer group.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80 years old
* Grade 2 or 3 hallux rigidus based on Coughlin and Shurnas classification
* Presence of good bone stock as determined on pre-operative x-rays not requiring bone grafting
* Capable of consenting for self

Exclusion Criteria:

* Patients <18 years of age
* Grade 1 or 4 hallux rigidus based on Coughlin and Shurnas classification
* Active bacterial infection of the foot
* Previous bilateral total knee arthroplasty
* Previous fracture or significant trauma to the ipsilateral knee
* Inflammatory anthropathy
* Gout
* Inadequate bone stock
* Previous anthrodesis or arthroplasty performed on the ipsilateral first MTP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | 2 years
  Pre-operative and post-operative clinical range of motion of the first MTP joint
Patient's Pain Level | 2 years
  Pre-operative and post-operative visual analog pain scale

SECONDARY OUTCOMES:
Patient's Quality of Life | 2 years
  Foot and Ankle Ability Measure (FAAM) sports score uses patient-report to determine function
Clinically-Assessed Foot and Ankle Function | 2 years
  American Orthopedic Foot and Ankle Score (AOFAS) Hallux Metatarsophalangeal-Interphalangeal Scale
Health Status | 2 years
  12-item short form health survey, use of concomitant medications, and changes in health status
Surgical Complications | 2 years
  Fractures, nerve injuries, blood loss, infection, etc.
Implant Failure | 2 years
  Failure of the Cartiva Synthetic Cartilage Implant
Secondary Surgical Intervention | 2 years
  Additional subsequent procedures, including removal, reoperation, revision, or supplemental fixation

CONTACTS AND LOCATIONS:
Overall Officials: Amgad Amin, MD, Principal Investigator — Department of Orthopedic Surgery and Rehabilitation

IPD SHARING:
Plan to Share IPD: No